CLINICAL TRIAL: NCT01685567
Title: INVESTIGATION of FLOW ALTERED, SHORT TRANSCERVICAL CAROTID ARTERY STENTING in PATIENTS With SIGNIFICANT CAROTID ARTERY DISEASE With Filter.
Brief Title: Safety and Efficacy Study for Reverse Flow Used During Carotid Artery Stenting Procedure
Acronym: ROADSTER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Silk Road Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SRM-2012-02
Record Dates: First submitted 2012-09-10; First posted 2012-09-14 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Carotid Artery Disease
Keywords: carotid artery disease; reverse flow
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MICHI NPS+f (Experimental): The MICHI™ NPS+f is a flow reversal circuit consisting of two proprietary sheaths connected by standard surgical tubing. The sheaths each have a standard hemostasis valve and sidearm. An in-line flow regulator allows the clinician to modify to the flow through the circuit (either high flow or low flow) in addition to permitting temporary cessation of flow.
  Interventions: Device: MICHI NPS+f

INTERVENTIONS:
Device: MICHI NPS+f — Cerebral protection with carotid flow reversal
  Other Names: ENROUTE Transcarotid Neuroprotection System

SUMMARY:
The purpose of this study is to obtain and establish the safety and efficacy of The MICHI™ Neuroprotection System with Filter (MICHI™ NPS+f) for providing cerebral embolic protection during angioplasty and stenting procedures in carotid arteries. The MICHI NPS+f also facilitates access to the carotid and neuro anatomy for the introduction of therapeutic or diagnostic endovascular devices and/or agents. It will be used in conjunction with a FDA approved carotid artery stent for the treatment of carotid artery disease.

DETAILED DESCRIPTION:
Cerebral embolization during carotid artery stenting (CAS) can often precipitate severe adverse neurological effects. Most major clinical studies of CAS have used distal filters for cerebral protection and have compared the neurologic complication rates with those of carotid endarterectomy (CEA). Many currently available embolic protection devices, however, have limited efficacy in capturing microembolic debris that is liberated during stenting, pre-dilatation and post-dilatation. Distal protection systems are furthermore limited by the need to cross the lesion prior to deployment. Some studies have shown a relatively high incidence of cerebral infarction even when distal protection devices are employed.

Cerebral protection with carotid flow reversal is a method that was developed as an alternative to the use of distal protection devices. While novel in its approach, this method too has its limitations. Another technique developed employs carotid flow reversal prior to traversing the stenosis and can be accomplished by directly accessing the carotid anatomy without the use of the transfemoral approach. Major benefits to this method include a simpler route to the target lesion and the ability to perform the procedure on patients with severe carotid tortuosity and difficult aortic arch anatomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must meet one of the following criteria regarding neurological symptom status and degree of stenosis:

   * Symptomatic: Stenosis must be greater than or equal to 50% as determined by angiogram and the patient has a history of stroke (minor or non-disabling), TIA and/or amaurosis fugax within 180 days of the procedure.
   * Asymptomatic: Stenosis must be greater than or equal to 70% as determined by angiogram without any neurological symptoms within the prior 180 days.
2. Target vessel must meet diameter requirements for stent (refer to selected stent IFU for diameter requirements).
3. Patient has a discrete lesion located in the internal carotid artery (ICA) with or without involvement of the contiguous common carotid artery (CCA).
4. Patient is greater or equal to 18 years of age.
5. Patient has no childbearing potential or has a negative pregnancy test within one week prior to the study procedure.
6. Patient understands the nature of the procedure and has provided a signed informed consent using a form that has been reviewed and approved by the Investigational Review Board/Ethics Committee of the respective clinical site prior to the procedure. This will be obtained prior to participation in the study.
7. Patient is willing to comply with the protocol requirements and return to the treatment center for all required clinical evaluations.
8. Patient meets at least one of the anatomic or clinical high-risk criteria.

Exclusion Criteria:

1. Patient has chronic atrial fibrillation.
2. Patient has had any episode of paroxysmal atrial fibrillation within the past 6 months, or history of paroxysmal atrial fibrillation requiring chronic anticoagulation.
3. Patient has an evolving stroke.
4. Patient has severe dementia.
5. Patient has a history of spontaneous intracranial hemorrhage within the past 12 months.
6. Patient has had a recent (<7 days) stroke of sufficient size (on CT or MRI) to place him or her at risk of hemorrhagic conversion during the procedure.
7. Patient had hemorrhagic transformation of an ischemic stroke within the past 60 days.
8. Patient has active bleeding diathesis or coagulopathy or will refuse blood transfusion.
9. Patient had or will have CABG, endovascular stent procedure, valve intervention or vascular surgery within 30 days before or after the intervention.
10. Patient has had a recent GI bleed that would interfere with antiplatelet therapy.
11. Life expectancy of < 12 months post procedure.
12. Patient has history of intolerance or allergic reaction to any of the study medications or stent materials (refer to stent IFU), including aspirin (ASA), ticlopidine, clopidogrel, prasugrel, statin or contrast media (that can't be pre medicated). Patients must be able to tolerate statins and a combination of ASA and ticlopidine, ASA and clopidogrel or ASA and prasugrel.
13. Myocardial Infarction within 72 hours prior to the intervention.
14. Presence of a previous placed intravascular stent in target vessel or the planned arteriotomy site.
15. Patient has had neurologic illnesses within the past two years characterized by fleeting or fixed neurologic deficit which cannot be distinguished from TIA or stroke (e.g. partial or secondarily generalized seizures, complicated or classic migraine, tumor or other space-occupying brain lesions, subdural hematoma, cerebral contusion or other post-traumatic lesions, intracranial infection, demyelinating disease, moderate to severe dementia, or intracranial hemorrhage).
16. Patient with a history of major stroke (CVA or retinal embolus) with major neurological deficit likely to confound study endpoints within 1 month of index procedure.
17. Patient has Hgb <10 g/dl, platelet count <125,000/μl, uncorrected INR >1.5, bleeding time >1 minute beyond upper limit normal, or heparin-associated thrombocytopenia.
18. Patient has an intracranial tumor.
19. Patient is actively participating in another drug or device trial (IND or IDE) that has not completed the required protocol follow-up period.
20. Patient has inability to understand and cooperate with study procedures or provide informed consent.
21. Occlusion or [Thrombolysis In Myocardial Infarction Trial (TIMI 0)] "string sign" >1cm of the ipsilateral common or internal carotid artery.
22. Patient has vertebrobasilar insufficiency symptoms only, without clearly identifiable symptoms referable to the study carotid artery.
23. Knowledge of cardiac sources of emboli.e.g. left ventricular aneurysm, intracardiac filling defect, cardiomyopathy, aortic or mitral prosthetic heart valve, calcific aortic stenosis, endocarditis, mitral stenosis, atrial septal defect, atrial septal aneurysm, or left atrial myxoma).
24. Recently (<60 days) implanted heart valve (either surgically or endovascularly), which is a known source of emboli as confirmed on echocardiogram.
25. Ostium of Common Carotid Artery (CCA) requires revascularization.
26. Presence of extensive or diffuse atherosclerotic disease involving the proximal common carotid artery that would preclude the safe introduction of the study device.
27. The patient has less than 5cm between the clavicle and bifurcation, as assessed by duplex Doppler ultrasound.
28. Bilateral carotid stenosis if intervention is planned within 37 days of the index procedure.
29. An intraluminal filling defect (defined as an endoluminal lucency surrounded by contrast, seen in multiple angiographic projections, in the absence of angiographic evidence of calcification) that is not associated with an ulcerated target lesion.
30. Abnormal angiographic findings: ipsilateral intracranial or extracranial arterial stenosis greater in severity than the lesion to be treated, cerebral aneurysm > 5 mm, AVM (arteriovenous malformation) of the cerebral vasculature, or other abnormal angiographic findings.
31. Patient has had a previous intervention in the ipsilateral proximal CCA.
32. Patient has had a TIA or amaurosis fugax within 48 hours prior to the procedure.
33. Patient has contralateral lateral recurrent, laryngeal or vagus nerve injury.
34. Patient is otherwise unsuitable for intervention in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2012-11; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Kwolek, MD, Principal Investigator — Massachusetts General Hospital; Richard Cambria, MD, Principal Investigator — Massachusetts General Hospital
Locations (21):
- United States (20):
  - Peter Morton UCLA Medical Center, Los Angeles, California
  - Florida Hospital, Orlando, Florida
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - McLaren Regional Medical Center, Flint, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Albany Medical Center, Albany, New York
  - University at Buffalo Neurosurgery, Inc, Buffalo, New York
  - Columbia University, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University Hospitals Case Medical Center and Case Western Reserve University School of Medicine, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Jobst Vascular Institute, Toledo, Ohio
  - Oklahoma Heart, Oklahoma City, Oklahoma
  - Greenville Hospital System, Greenville, South Carolina
  - Cardiothoracic & Vascular Surgeons, Austin, Texas
  - Methodist Medical Center, Dallas, Texas
  - Dallas VA Medical Center, Dallas, Texas
  - Sentara Vascular Specialists, Norfolk, Virginia
- Hospital Virgen de la Salud, Toledo, Spain

REFERENCES:
- [Result] Kwolek CJ, Jaff MR, Leal JI, Hopkins LN, Shah RM, Hanover TM, Macdonald S, Cambria RP. Results of the ROADSTER multicenter trial of transcarotid stenting with dynamic flow reversal. J Vasc Surg. 2015 Nov;62(5):1227-34. doi: 10.1016/j.jvs.2015.04.460. PMID 26506270
- [Result] Alpaslan A, Wintermark M, Pinter L, Macdonald S, Ruedy R, Kolvenbach R. Transcarotid Artery Revascularization With Flow Reversal. J Endovasc Ther. 2017 Apr;24(2):265-270. doi: 10.1177/1526602817693607. Epub 2017 Feb 17. PMID 28335706
- [Derived] Chung J, Kumins NH, Smith J, Motaganahalli RL, Schneider PA, Kwolek CJ, Kashyap VS; ROADSTER Investigators. Physiologic risk factors increase risk of myocardial infarction with transcarotid artery revascularization in prospective trials. J Vasc Surg. 2023 Apr;77(4):1192-1198. doi: 10.1016/j.jvs.2022.12.013. Epub 2022 Dec 20. PMID 36563712
- [Derived] Malas MB, Leal Lorenzo JI, Nejim B, Hanover TM, Mehta M, Kashyap V, Kwolek CJ, Cambria R. Analysis of the ROADSTER pivotal and extended-access cohorts shows excellent 1-year durability of transcarotid stenting with dynamic flow reversal. J Vasc Surg. 2019 Jun;69(6):1786-1796. doi: 10.1016/j.jvs.2018.08.179. Epub 2019 Jan 2. PMID 30611582
- See also: Results of the ROADSTER multicenter trial of transcarotid stenting with dynamic flow reversal. — https://www.ncbi.nlm.nih.gov/pubmed/?term=26506270
- See also: Transcarotid Artery Revascularization with Flow Reversal: the PROOF Study — https://www.ncbi.nlm.nih.gov/pubmed/28335706

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment opened November, 2012 and ended March, 2016.
Groups:
- Intention-to-Treat (ITT): All patients who were enrolled in the pivotal phase of the study are included. Lead-in patients are not included in this group.
Period: Overall Study
Arm/Group | Intention-to-Treat (ITT)
Started | 219
Completed | 219
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intention-to-Treat (ITT)
Number analyzed (Participants) | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.30 (8.574)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 136
Symptomatic Status [Count of Participants; unit: Participants]
  Asymptomatic | 175
  Symptomatic | 44

OUTCOME MEASURES:

1. Primary Outcome: Hierarchical Composite of Stroke, Myocardial Infarction, and Death
Description: The primary endpoint was a hierarchical composite of any stroke, myocardial infarction and death during a 30-day post-procedural period in the ITT (pivotal and extended enrollment) population comprised of subjects deemed to be high risk for complications from CEA.
Time Frame: 30-day post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intention-to-Treat (ITT)
Number analyzed (Participants) | 219
Participants | 8

2. Secondary Outcome: All Death (Non-hierarchical)
Description: The analyses to be conducted on the secondary endpoints are intended to provide additional supportive evidence of the efficacy and safety of the device.
Time Frame: 0 to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intention-to-Treat (ITT)
Number analyzed (Participants) | 219
Participants | 2

3. Secondary Outcome: All Myocardial Infarctions (Non-hierarchical)
Description: as for outcome 2
Time Frame: 0 to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intention-to-Treat (ITT)
Number analyzed (Participants) | 219
Participants | 4

4. Secondary Outcome: All Stroke (Non-hierarchical)
Description: as for outcome 2
Time Frame: 0 to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intention-to-Treat (ITT)
Number analyzed (Participants) | 219
Participants | 2

5. Secondary Outcome: Ipsilateral Stroke (Non-hierarchical)
Description: Data on ipsilateral stroke 31-365 days post procedure will be collected to provide additional supportive evidence of the safety of the device.
Time Frame: 31-365 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intention-to-Treat (ITT)
Number analyzed (Participants) | 219
Participants | 3

ADVERSE EVENTS:
Arm/Group | Intention-to-Treat (ITT)
Serious Adverse Events (participants affected / at risk) | 29/219
Other Adverse Events (participants affected / at risk) | 118/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intention-to-Treat (ITT) (N=219)
Anaemia (Blood and lymphatic system disorders) | 5
Myocardial Infarction (Cardiac disorders) | 3
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Pneumonia (Infections and infestations) | 2
Wound Haematoma (Injury, poisoning and procedural complications) | 3
Angina Pectoris (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 1
Cardiac Failure Acute (Cardiac disorders) | 1
Post Procedural Cellulitis (Infections and infestations) | 1
Incision Site Haematoma (Injury, poisoning and procedural complications) | 2
Troponin Increased (Investigations) | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Ischaemic Stroke (Nervous system disorders) | 1
Metabolic Encephalopathy (Nervous system disorders) | 1
Psychomotor Seizures (Nervous system disorders) | 1
Renal Failure (Renal and urinary disorders) | 2
Urinary Retention (Renal and urinary disorders) | 2
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Aortic Aneurysm (Vascular disorders) | 1
Artery Dissection (Vascular disorders) | 4
Hypotension (Vascular disorders) | 4
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intention-to-Treat (ITT) (N=219)
Anaemia (Blood and lymphatic system disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Angina Pectoris (Cardiac disorders) | 2
Atrial Fibrillation (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 5
Cardiac Arrest (Cardiac disorders) | 1
Cardiac Failure Acute (Cardiac disorders) | 1
Myocardial Infarction (Cardiac disorders) | 4
Sinus Bradycardia (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 1
Ventricular Extrasystoles (Cardiac disorders) | 1
Ear Pain (Ear and labyrinth disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 3
Chest Discomfort (General disorders) | 1
Device Occlusion (General disorders) | 1
Oedema (General disorders) | 1
Pain (General disorders) | 25
Pyrexia (General disorders) | 9
Vessel Puncture Site Haematoma (General disorders) | 4
Allergy To Arthropod Bite (Immune system disorders) | 1
Acute Sinusitis (Infections and infestations) | 1
Adenoviral Upper Respiratory Infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Herpes Zoster (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Post Procedural Cellulitis (Infections and infestations) | 1
Rash Pustular (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 4
Cranial Nerve Injury (Injury, poisoning and procedural complications) | 1
Incision Site Haematoma (Injury, poisoning and procedural complications) | 4
Vascular Injury (Injury, poisoning and procedural complications) | 1
Wound Haematoma (Injury, poisoning and procedural complications) | 7
Wound Secretion (Injury, poisoning and procedural complications) | 8
Blood Creatine Phosphokinase Increased (Investigations) | 3
Oxygen Saturation Decreased (Investigations) | 1
Troponin Increased (Investigations) | 7
Dehydration (Metabolism and nutrition disorders) | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypokalaemic Syndrome (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Carotid Artery Stenosis (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Ischaemic Stroke (Nervous system disorders) | 1
Metabolic Encephalopathy (Nervous system disorders) | 1
Psychomotor Seizures (Nervous system disorders) | 1
Hallucination, Visual (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 4
Renal Failure (Renal and urinary disorders) | 2
Urinary Retention (Renal and urinary disorders) | 11
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Skin Irritation (Skin and subcutaneous tissue disorders) | 1
Therapy Regimen Changed (Surgical and medical procedures) | 1
Aortic Aneurysm (Vascular disorders) | 1
Artery Dissection (Vascular disorders) | 9
Hemorrhage (Vascular disorders) | 1
Hematoma (Vascular disorders) | 1
Hypertension (Vascular disorders) | 9
Hypotension (Vascular disorders) | 23
Orthostatic Hypotension (Vascular disorders) | 2
Vascular Occlusion (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No